CLINICAL TRIAL: NCT04899635
Title: Profiling Biomechanical Responses and Workload of the Human Myocardium to Explore the Concept of Myocardial Fatigue and Reversibility
Brief Title: POWER Myocardial Fatigue Study: a Biomechanical Assessment of Contractility of Human Myocardium
Acronym: POWER
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Coventry University (Other)
Responsible Party: Sponsor
Other Study IDs: PB528721
Record Dates: First submitted 2021-05-11; First posted 2021-05-24 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure; Fatigue; Muscle, Heart; Myocardial Dysfunction; Exhaustion; Heart
Keywords: Myocardial Fatigue; Preload; Afterload; Cardiac Work-loop; Cardiomyocytes; Biomechanical model
MeSH Terms: conditions — Heart Failure; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diseased cardiac tissue: Heart muscle or cells (cardiomyocytes) will be obtained from patients undergoing cardiac surgery, namely coronary artery bypass grafting or for severe valvular heart disease.
  Interventions: Other: In-vitro contractile fatigue protocol
- Healthy cardiac tissue: Healthy donor hearts from deceased individuals that are not transplantable due to technical reasons
  Interventions: Other: In-vitro contractile fatigue protocol

INTERVENTIONS:
Other: In-vitro contractile fatigue protocol — Using contractility assays for muscle slices or the work-loop assay for isolated heart cells, the tissue preparation will undergo a series of contraction and relaxation under varying levels of preload, afterload, stimulation frequency and under other experimental conditions such as drug-induced inotropism.

SUMMARY:
To gain a comprehensive understanding of the biomechanical behaviour of human heart to explore the concept of myocardial fatigue in response to a temporal range of preload, afterload and drug-induced inotropy using in-vitro contractile assays.

DETAILED DESCRIPTION:
A continuum of pathological states from fatigue, injury to damage of the myocardium has been proposed which complements the continuous spectrum of HF and reconciles the seemingly disparate plethora of mechanisms behind the pathophysiology of HF. Unlike skeletal muscle where mechanical stress can be readily removed upon fatigue, an impaired left ventricle continues to receive preload from the right ventricle and cannot rest, maintaining cardiac output only at the expense of increasing filling pressures (as in HF with preserved ejection fraction). If concurrently faced with high afterload from vascular stiffness, ventricular-arterial decoupling occurs, driving mechanical inefficiency and diminishing cardiac output (as in HF with reduced ejection fraction). Chances of recovery is linked to the degree of fatigue, cardiomyocyte loss and replacement with non-contractile fibrosis. Assuming that the myocardium is in a state of chronic fatigue before reaching advanced stages of fibrosis, cases such as aortic stenosis or hypertensive heart disease may potentially be reversible if the pathological load is promptly removed.

This study will be re-synthesizing existing knowledge of the biomechanical behaviour of healthy and diseased cardiac myocytes and muscle in a new light of the theoretical constructs of myocardial fatigue, aligned with the existing energy-starvation theory. It will be a proof-of-concept study. Just as Frank-Starling's relationship between preload and cardiac output emerged from pre-clinical studies on muscle behaviour with subsequently major clinical implications, this study represents a necessary stepping stone to adding a new layer of insight into the pathophysiology of heart failure (HF).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients between 18 to 85-years old undergoing open-heart surgery who can undergo the consent process for the study
* Healthy donor hearts that are deemed non-transplantable and consent received from a legal representative

Exclusion Criteria:

This criterion is kept to a minimum since the availability of human myocardial samples is finite and dependent on the limited number of patients undergoing cardiac surgery annually within the local hospital.

* Patients who do not have the mental capacity to undergo the consent process
* For the safety of researchers, patients with evidence of ongoing blood-borne infections such as HIV, or a recent positive test for COVID-19 (within 10 days of last PCR test).

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Human cardiac tissues (atrial appendages and ventricular tissue biopsies) are obtained from patients undergoing elective or inpatient open-heart surgery, namely coronary artery bypass grafting and valvular replacement. If available, explanted failing hearts are also recruited for experimentation. A control population consists of healthy donor hearts that are deemed non-transplantable and collected by the Arden Tissue Bank at UHCW.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the force generated by the muscle cell and/or muscle slice | Within a day for each experiment
  This will be based on the effects of changing load and/or exposure to drug-induced inotropic effects
Changes in the velocity of shortening by the muscle cell and/or muscle slice | Within a day for each experiment
  This will be based on the effects of changing load and/or exposure to drug-induced inotropic effects
Changes in the end-systolic force-length relationship of the muscle cell and/or muscle slice | Within a day for each experiment
  This will be based on the effects of changing load and/or exposure to drug-induced inotropic effects, and calculated by integrating the above force and length changes.

SECONDARY OUTCOMES:
Changes in the phosphorylation potential | Within a day for each experiment
  This will be calculated by determining the above concentration of adenosine triphosphate and its metabolic by-product including inorganic phosphate, at different times of the contraction fatigue protocol (e.g. before, during, and after).
Changes in the phosphocreatine/ATP ratio | Within a day for each experiment
  This will be calculated by determining the above concentration of phosphocreatine and ATP at different times of the contraction fatigue protocol (e.g. before, during and after).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry and Warwickshire, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tran P, Joshi M, Banerjee P. Concept of myocardial fatigue in reversible severe left ventricular systolic dysfunction from afterload mismatch: a case series. Eur Heart J Case Rep. 2021 Mar 7;5(3):ytab089. doi: 10.1093/ehjcr/ytab089. eCollection 2021 Mar. PMID 34113768
- [Background] Banerjee P. Heart failure: a story of damage, fatigue and injury? Open Heart. 2017 Oct 15;4(2):e000684. doi: 10.1136/openhrt-2017-000684. eCollection 2017. PMID 29081980